CLINICAL TRIAL: NCT03429101
Title: A Phase 1b Study of Poziotinib in Combination With T-DM1 in Women With Advanced or Metastatic HER2-Positive Breast Cancer
Brief Title: A Study of Poziotinib in Combination With T-DM1 in HER2-Positive Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose limiting toxicity
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-101
Record Dates: First submitted 2018-01-18; First posted 2018-02-12 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Poziotinib; HER2 Positive; T-DM1
MeSH Terms: conditions — Breast Neoplasms | interventions — HM781-36B; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Intervention Model Description: * Part 1: Dose Finding To determine the MTD/MAD of poziotinib in combination with the standard dose of T-DM1 by using a "3+3" design. At least 3 patients may be enrolled in each cohort before a decision is made to proceed to the next cohort.
  * Part 2: MTD/MAD Expansion An additional 10 patients will be treated at the dose identified during Part 1 of the study to further evaluate the safety and efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Poziotinib (Experimental): * Part 1: Dose Finding The MTD/MAD of poziotinib in combination with the standard dose of T-DM1 will be determined by using a "3+3" design. At least 3 patients may be enrolled in each cohort before a decision is made to proceed to the next cohort.
  * Part 2: MTD/MAD Expansion An additional 10 patients will be treated at the dose identified during Part 1 to further evaluate the combination at the MTD or the MAD.
  Interventions: Drug: Poziotinib; Drug: T-DM1

INTERVENTIONS:
Drug: Poziotinib — Poziotinib is a tablet for oral administration.
Drug: T-DM1 — T-DM1 (ado-trastuzumab emtansine) is a HER2-targeted therapy for I.V. administration.
  Other Names: ado-trastuzumab emtansine

SUMMARY:
This is a Phase 1b, open-label, multicenter study to determine the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of poziotinib when administered with standard dosing of T-DM1 (3.6 mg/kg IV on Day 1 of each 21-day cycle) in women with advanced or metastatic HER2+ breast cancer. The poziotinib dose identified in Part 1 of the study will be used in combination with standard dose of T-DM1 in Part 2 of the study to confirm the poziotinib dose and evaluate the preliminary efficacy of the combination therapy.

DETAILED DESCRIPTION:
In Part 1, the dose of poziotinib, in combination with the standard dose of T-DM1 (3.6 mg/kg IV) on Day 1 of each cycle will be determined using a "3+3" design with up to 3 dose levels tested beginning with 8 mg/day.

Poziotinib dose escalation/de-escalation for the next dose cohort will proceed based on the occurrence of dose-limiting toxicities (DLTs) during Cycle 1 of the dose cohort. Patients in the dose cohort, if not discontinued, will continue treatment until discontinuation.

In Part 2 of the study, approximately 10 patients will be treated at the MTD/MAD to confirm dose for safety of the combination and to evaluate preliminary efficacy. Treatment for all patients will continue until disease progression, unacceptable toxicity, or continuation of study treatment is not in the best interest of the patient.

The Screening period (Day -30 to Day -1) will last up to 30 days prior to Cycle 1, Day 1.

During each 21-day cycle, eligible patients will receive poziotinib at the assigned dose, orally, once daily. T-DM1 3.6 mg/kg IV will be administered on Day 1 of each treatment cycle.

All treated patients will be followed for response until disease progression or the start of new treatment and then for survival (3 year study duration).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be female, at least 18 years of age, but not older than 90 years, with advanced or metastatic HER2+ breast cancer and a life expectancy of more than 6 months
* Patient must have confirmed HER2 overexpression or gene-amplified tumor via immunohistochemistry [IHC] with IHC 3+ or IHC 2+ with confirmatory fluorescence in situ hybridization [FISH]+ or [ISH]+
* Patients must have had at least 1 line of anti-HER2 directed therapy either in the metastatic or early-stage disease setting
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Patient has had previous treatment with poziotinib.
* Patient has received anticancer chemotherapy, TKIs, biologics, immunotherapy, radiotherapy, or investigational treatment within 15 days. (There is no washout for hormonal therapy for breast cancer).
* Patient has a life expectancy less than 3 years due to other malignancies.
* Patient is pregnant or breast-feeding.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3 Years
  Evaluate the Objective Response Rate (ORR) in patients treated with daily poziotinib in combination with T-DM1 (every 3 weeks) in women with advanced or metastatic HER2 positive breast cancer.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 27 weeks
  Evaluate the Disease Control Rate (DCR) at 9, 18, and 27 weeks in patients treated at the MTD/MAD.
Progression-free Survival (PFS) | 3 years
  Evaluate Progression-free Survival (PFS) in patients treated with MTD/MAD.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Los Angeles Hematology Oncology Medical Group, Glendale, California